CLINICAL TRIAL: NCT03905460
Title: Point-of-care Ultrasound in Prehospital Dyspnea: Game-changer or Gaming-gadgets?
Brief Title: Point-of-care Ultrasound in Prehospital Dyspnea
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Morten Thingemann Bøtker, Associate Professor, University of Aarhus
Other Study IDs: POC Ultrasound
Record Dates: First submitted 2019-03-21; First posted 2019-04-05 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound — Focused ultrasound of the heart, lungs and pleurae

SUMMARY:
Point-of-care ultrasound in patients with dyspnoea has been shown to alter patient treatment and the time to correct treatment when performed in emergency departments. In Denmark, physician-staffed ambulances are sent to citizens with severe ABCD symptoms including dyspnoea. Hence, there is a potential for correct diagnostics and appropriate treatment already in the citizens' own home or en route to the hospital. This study aims to evaluate the clinical performance of prehospital point-of-care ultrasound in patients with dyspnoea.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 18 years
* dyspnea as a dominating complaint At least one of
* respiratory frequency >25/minute
* oxygen saturation < 95%
* oxygen therapy initiated

Exclusion Criteria:

* trama patients
* prior enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All citizens who have contacted the Acute Medical Coordination center in the Central Denmark Region for emergency medical treatment.
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity for diagnosing heart failure | From initial citizen contact to end of ultrasound examination within 15 minutes
  Change in sensitivity for diagnosing heart failure when adding point-of-care ultrasound to the clinical examination

SECONDARY OUTCOMES:
Sensitivity, clinical exam | From initial citizen contact and within a time-span of 15 minutes
  Sensitivity of clinical examination for for diagnosing heart failure. Held up against a post-hoc expert panel statement.
Sensitivity, Ultrasound examination | From initial citizen contact and within a time-span of 15 minutes
  Sensitivity of clinical examination supplemented with ultrasound scan for diagnosing heart failure. Held up against a post-hoc expert panel statement.
Treatment changes in medicine caused by ultrasound examination | From initial citizen contact and within a time-span of 15 minutes
  Changes in medical treatment including diuretics, nitric oxide, bronkodilation and steroids caused by the addition of an ultrasound scan
Treatment changes in ventilation caused by ultrasound examination | From initial citizen contact and within a time-span of 15 minutes
  Treatment changes ventilatory strategy including nasal cannula oxygen therapi, face mask or non-invasive positive pressure ventilation caused by the addition of an ultrasound scan
Triage changes caused by ultrasound examination | From initial citizen contact and within a time-span of 60 minutes
  Change in the department or hospital that the patient is sent to as a cause of an ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bøtker, MD, Phd, Principal Investigator — Prehospital of Central Denmark Region
Locations (1):
- Præhospitalet, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gundersen EA, Juhl-Olsen P, Bach A, Rostgaard-Knudsen M, Nielsen BRR, Skaarup SH, Petersen HO, Fjolner J, Poulsen MGG, Botker MT. PrehospitaL Ultrasound in Undifferentiated DyspnEa (PreLUDE): a prospective, clinical, observational study. Scand J Trauma Resusc Emerg Med. 2023 Feb 5;31(1):6. doi: 10.1186/s13049-023-01070-4. PMID 36740691